CLINICAL TRIAL: NCT00949572
Title: Characterisation of Human Disseminated Cellular and Humoral Immune Responses Following Sublingual or Intramuscular Deposition of Antigens
Brief Title: Measuring Responses to Sublingual Antigens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: European Union (Other)
Responsible Party: David J.M. Lewis / Principal Investigator, St George's, University of London
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SG09-EN01; REC number: 09/80803/77 (Other: NRES, UK); EC grant number 201038 (Other: European Commission)
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Sexually Transmitted Diseases, Viral
Keywords: mucosal immunity; immunization; sublingual
MeSH Terms: conditions — Sexually Transmitted Diseases, Viral | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intramuscular administration (Experimental): Intramuscular injection of HPV vaccine proteins
  Interventions: Biological: Human Papillomavirus 6,11,16,18 Vaccine Recombinant alum ads
- Sublingual administration (Experimental): Sublingual administration of HPV vaccine proteins
  Interventions: Biological: Human Papillomavirus 6,11,16,18 Vaccine Recombinant alum ads

INTERVENTIONS:
Biological: Human Papillomavirus 6,11,16,18 Vaccine Recombinant alum ads — 1 intramuscular dose (0.5 ml) on month 0, 1 and 4 containing approximately: Human Papillomavirus Type 6 L1 protein 20 micrograms Human Papillomavirus Type 11 L1 protein 40 micrograms Human Papillomavirus Type 16 L1 protein 40 micrograms Human Papillomavirus Type 18 L1 protein 20 micrograms
  Other Names: Gardasil
  Arms: Intramuscular administration
Biological: Human Papillomavirus 6,11,16,18 Vaccine Recombinant alum ads — 1 sublingual application on month 0, 1 and 4 of 0.5 ml containing approximately: Human Papillomavirus Type 6 L1 protein 20 micrograms Human Papillomavirus Type 11 L1 protein 40 micrograms Human Papillomavirus Type 16 L1 protein 40 micrograms Human Papillomavirus Type 18 L1 protein 20 micrograms
  Other Names: Gardasil
  Arms: Sublingual administration

SUMMARY:
This study is a preliminary investigation of immune responses, in the blood and in cervical & vaginal secretions, to proteins ("antigens") taken up across the undersurface of the tongue.

DETAILED DESCRIPTION:
Animal studies have shown that this "sublingual" surface can take up antigens and stimulate immune responses, which may have a different character to responses induced by injecting the same antigens. In previous studies of nasal and oral delivery, we used licensed vaccine preparations as pure and well-characterised model antigens safe for use in humans. We will use a licensed "HPV" vaccine as the source of antigens in this study. The quantity and character of responses (lymphocyte number and pattern of surface proteins, concentration and type of antibodies in fluids) will be measured in detail in various anatomical sites (blood, vaginal secretions) before and after delivery of antigens on three occasions. As well as using established immune assays to characterise the responses, we will develop new research assays to detect populations of lymphocytes and antibodies present in secretions. To ensure we have positive samples to include in our assays and validate new techniques, we will recruit some subjects to receive a standard intramuscular injection, as this is known to be nearly 100% reliable in inducing measurable immune responses. As this is a preliminary study we will recruit enough subjects (based on our previous experience with nasal, oral and injected delivery) to ensure we generate sufficient responses we can measure. We may be able to draw some tentative conclusions about differences in character of immune responses following sublingual or injected delivery, but it is not the intention of this initial study to formally compare these two routes. If we observe that sublingual delivery in humans can induce immune responses, we can select assays to test any differences more formally in subsequent bigger and more focused studies.

ELIGIBILITY:
Inclusion Criteria:

* A female adult volunteer aged between 18 and 35 years old.
* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Provide written informed consent following a detailed written explanation of participation in the protocol.
* They are in good health as determined by medical history, physical examination, haematology testing, and clinical judgement before entering into the study.
* They are available for the whole duration of the study.
* If of childbearing potential, must have a negative pregnancy test before each immunisation.
* They have not donated blood during 3 months prior to study entry and agree to not donate for 3 months after the end of their participation in the study.
* They are eligible for free medical treatment

Exclusion Criteria:

* They have already been vaccinated with an HPV vaccine
* They have participated in a clinical trial in the last 6 months in which they have been exposed to an investigational product (pharmaceutical product or placebo or device) or concurrent participation in another clinical research study at the time of enrolment.
* Use of any investigational or non-registered product (drug or vaccine) within 30 days preceding the first dose of challenge agent, or planned use during the study period.
* They are pregnant or breast-feeding.
* They have a known or suspected ongoing cervico-vaginal disease, malignancy or abnormality discovered at time of screening.
* They present in the samples obtained at the screening visit: positive results for HIV, HBs Ag, anti-HBc and anti-HCV antibody, a clinically significant abnormality in haematology. Normal ranges will be defined by the pathology laboratory undertaking assays.
* They have a clinically significant acute or chronic pulmonary, cardiovascular, hepatic or renal functional abnormality, blood or neurological disorders, immune dysfunction, autoimmune diseases, diabetes (excluding history of gestational diabetes), or malignancy at the time of enrolment, as determined by medical history, physical examination or laboratory screening tests.
* They have received any form of immunosuppressive therapy in the past 6 months.
* They are receiving any medications via vaginal route (as this may interfere with collection of samples).
* They have any tongue or frenulum piercings or oral jewellery that may interfere with sublingual delivery.
* They have received blood products or immunoglobulins 120 days prior to enrolment.
* They have thrombocytopaenia or any coagulation disorder (because bleeding may occur following an intramuscular administration in these individuals).
* Any other medical, psychiatric or social condition, drug treatment, occupational or other responsibility that, in the judgement of the investigator, would interfere with or serve as a contradiction to adherence to the study protocol or ability to give informed consent.
* Individuals who cannot read or speak fluent English.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Concentration and isotype profile of antigen-specific antibody in cervico-vaginal secretions measured by ELISA and/or LUMINEX assay | 0, 1, 4 and 5 months after first immunization

SECONDARY OUTCOMES:
Concentration and isotype profile of antigen-specific antibody in serum measured by ELISA and/or LUMINEX assay | 0, 1, 4 & 5 months after first immunization
Frequency and isotype profile of antigen-specific antibody secreting cells in blood | 0 and 1 week after each immunization
Frequency and expression profile of mucosa-associated homing, memory and regulatory markers on antigen-specific T cells in blood in response to in vitro antigen stimulation | 0 and 4 weeks after each immunization
Profile of cytokine secretion by peripheral blood mononuclear cells in response to in vitro antigen stimulation measured by ELISA | 0 and 4 weeks after each immunization

CONTACTS AND LOCATIONS:
Overall Officials: David JM Lewis, MD, Principal Investigator — St George's, University of London
Locations (1):
- St George's Vaccine Institute, St George's University of London, London, England, United Kingdom

REFERENCES:
- [Derived] Huo Z, Bissett SL, Giemza R, Beddows S, Oeser C, Lewis DJ. Systemic and mucosal immune responses to sublingual or intramuscular human papilloma virus antigens in healthy female volunteers. PLoS One. 2012;7(3):e33736. doi: 10.1371/journal.pone.0033736. Epub 2012 Mar 16. PMID 22438987
- See also: Website of St George's Vaccine Institute — http://www.vaccine.ac.uk
- See also: Website of St George's University of London — http://www.sgul.ac.uk
- See also: European Commission EURONEUT41 funding body website — http://ec.europa.eu/research/health/infectious-diseases/poverty-diseases/projects/200_en.htm